CLINICAL TRIAL: NCT02964065
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase Ⅲ Trial on the Efficacy, Safety and Immunogenicity of Live-Attenuated Influenza Vaccine (LAIV)
Brief Title: A Trial on the Efficacy, Safety and Immunogenicity of Live-Attenuated Influenza Vaccine (LAIV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: Simoon Record Pharma Information Consulting Co., Ltd. (Industry); National Institutes for Food and Drug Control, China (Other); Baoding Municipal Center for Disease Control and Prevention, Hebei, P.R.China (Unknown); Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Maoming Municipal Center for Disease Control and Prevention, Guangdong, P.R.China (Unknown); Department of Medical Statistics, Fourth Military Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: F20160728
Record Dates: First submitted 2016-11-11; First posted 2016-11-15 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Influenza
Keywords: Influenza Vaccines; LAIV
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAIV (Experimental): a single dose of Live-Attenuated influenza Vaccine;Dose: 0.2 ml; Each dose contains not less than 6.9 lg EID50 of type A live attenuated influenza virus reassortants(H1N1 and H3N2), and not less than 6.4 lg EID50 of type B live attenuated influenza virus reassortants.
  Interventions: Biological: Live-Attenuated influenza Vaccine(LAIV)
- Placebo (Placebo Comparator): a single dose of Placebo. Inactivated placebo will be identical to LAIV in appearance, ingredients and concentrations, attenuated influenza virus free.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Live-Attenuated influenza Vaccine(LAIV)
  Arms: LAIV
Biological: Placebo
  Arms: Placebo

SUMMARY:
This study is a Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase Ⅲ Trial to evaluate the efficacy, safety and immunogenicity of a single dose of Live-Attenuated influenza Vaccine(LAIV) among healthy children and adolescents aged 3-17 years.

DETAILED DESCRIPTION:
This study is a Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase Ⅲ Trial to evaluate the efficacy, safety and immunogenicity of a single dose of Live-Attenuated influenza Vaccine(LAIV) among healthy children and adolescents aged 3-17 years old. The subjects will be randomized in a 1:1 ratio of LAIV to placebo. Each subject will be vaccinated with a single dose of LAIV or Placebo. For evaluation of efficacy, subjects meeting the protocol-defined clinical case definition the 14th day post-vaccination will have a nasal swab collected for testing by RT-PCR or virus culture for evidence of influenza virus infection. All adverse events will be collected 30 minutes, 0-30 days after vaccination and all serious adverse events during the entire trial period. Blood samples will be collected from a part of subjects before vaccination and at the 30th day after immunization. Serum samples will be centrifuged for detection of antibodies to H1N1, H3N2, and influenza B.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children and adolescents aged 3-17 years old.
2. Informed consent obtained and signed by subjects or legal guardians prior to screening. Children or adolescents aged 10-17 yrs need sign informed consent by themselves.
3. Willing to participate for the planned duration of the study, including availability for follow-up.

Exclusion Criteria:

1. Any investigational or unregistered product (drug, vaccine or device) was used within 30 days, or planned to be used during the trial.
2. have been vaccinated with any influenza vaccine within 6 months, or plan to be vaccinated during the trail.
3. Immunosuppressive agents or other immunomodulatory drugs (defined as continuous use for more than 14 days) were used over a 3-month period.
4. Immunoglobulins and / or any blood products were used within 3 months, or planned to be used before blood collection.
5. History of Guillain-Barré syndrome; History of hypersensitivity to any component of the LAIV, including egg or egg products.
6. Severe allergic reactions after vaccination (including anaphylactic shock, allergic laryngeal edema, allergic purpura, local allergic necrosis).
7. Acute diseases , infections or febrile diseases (axillary temperature ≥37.1℃) on the day of vaccination.
8. Obvious coagulation dysfunction or History of anticoagulant therapy
9. Aspirin is being used(Salicylates are a potential risk factor for Reye syndrome)
10. Known or suspected immune deficiency diseases or immunosuppressed
11. Heart disease, respiratory diseases (including severe rhinitis, nasal deformities, polyps, etc.), liver disease, kidney disease, mental disorders, chronic infections etc.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9000 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects With Symptomatic, Laboratory-confirmed(RT-PCR/ Virus Culture) Influenza Virus Infection(Vaccine-like Strains) | Through 2 weeks to 1 year post vaccination

SECONDARY OUTCOMES:
Percentage of Subjects With Symptomatic, Laboratory-confirmed(RT-PCR/ Virus Culture) Influenza Virus Infection(Regardless of Vaccine Match) | Through 2 weeks to 1 year post vaccination
Percentage of Subjects with influenza-like illness caused by Influenza Virus Infection(Laboratory-confirmed by RT-PCR/ Virus Culture) | Through 2 weeks to 1 year post vaccination
Adverse Events Occurring Within 30 Minutes of Administration of Study Vaccine | Through 30 minutes post vaccination
Solicited Adverse Events | Through 14 days post vaccination
Unsolicited Adverse Events | Through 30 days post vaccination
Serious Adverse Events | Through 1 year post vaccination
Geometric Mean Titers (GMT) of Hemagglutination Inhibition (HAI) Antibodies to each of the Influenza Strains in the Vaccine Received | 30 days post vaccination
Percentage of subjects with antibody positive conversion to each of the Influenza Strains in the Vaccine Received. | 30 days post vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Guangdong Provincial Institute of Biological Products and Materia Media, Guangzhou, Guangdong
  - Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei
  - Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ai L, Gao Z, Lv H, Zhang J, Xu N, Zhao H, Lu Q, Zhu H, Shi N, Wei W, Liu D, Yu Q. Immunogenicity and safety of live attenuated influenza vaccine in children aged 3-17 years in China. Vaccine. 2025 Feb 6;46:126653. doi: 10.1016/j.vaccine.2024.126653. Epub 2024 Dec 26. PMID 39729925
- [Derived] Wang S, Zheng Y, Jin X, Gan Z, Shao Y, Zhu C, Hu X, Liang Z, Chen Y, Xing B, Lv H, Xu N. Efficacy and safety of a live attenuated influenza vaccine in Chinese healthy children aged 3-17 years in one study center of a randomized, double-blind, placebo-controlled phase 3 clinical trial, 2016/17 season. Vaccine. 2020 Aug 27;38(38):5979-5986. doi: 10.1016/j.vaccine.2020.07.019. Epub 2020 Jul 31. PMID 32747213